CLINICAL TRIAL: NCT05334173
Title: Randomized Clinical Trial on the Outcome of Gastric Bypass With Biliopancreatic and Alimentary Limbs of 150 Centimeters (cm)/70 cm Versus(vs) 70/150 cm, Measuring the Length of the Common Limb
Brief Title: Gastric Bypass With Different Lengths of the Bilipancreatic Limb
Acronym: BPG-1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Principal Investigator, Débora Acín, MD, PhD, Bariatric Surgeon, Hospital Universitario de Fuenlabrada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPG-1
Record Dates: First submitted 2022-03-19; First posted 2022-04-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Laparoscopic-Roux-en-Y Gastric Bypass; Obesity; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Sleep Apnea
Keywords: Diabetes Mellitus, Type 2; Hypertension; Dyslipidemia; Obstructive Sleep Apnea Syndrome; Quality of life; Nutritional deficit; Laparoscopic-Roux-en-Y-Gastric-Bypass; Biliopancreatic limb; Alimentary limb; Common limb
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Randomized trial in blocks (1:1). Type 1 laparoscopic Gastric Bypass (150cm alimentary limb and 70cm biliopancreatic limb) or type 2 laparoscopic Gastric Bypass (70cm alimentary limb and 150cm biliopancreatic limb)
Who Masked: Participant
Masking Description: Blinded for the patient and to the surgeon up to the time of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB TYPE 1 - LONGER ALIMENTARY LIMB (LAL-GB) (Active Comparator): 150 cm alimentary limb and 70 cm biliopancreatic limb
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB) measuring the lengh of the common limb
- RYGB TYPE 2 - LONGER BILIOPANCREATIC LIMB (LBPL-GB) (Active Comparator): 70 cm alimentary limb and 150 cm biliopancreatic limb
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB) measuring the lengh of the common limb

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGB) measuring the lengh of the common limb — The patients are randomized to Type 1 laparoscopic RYGB (150cm alimentary limb and 70cm biliopancreatic limb) or type 2 laparoscopic RYGB (70cm alimentary limb and 150cm biliopancreatic limb). In both groups, the total intestinal length is measured to determine the size of the common limb. We introduce a 10 cm ruler into the abdominal cavity to measure the bowel and then extract it. LRYGB is made with linear stapler anastomosis.
  Other Names: Biliopancreatic and alimentary limbs of 150cm / 70cm; Biliopancreatic and alimentary limbs of 70cm / 150cm

SUMMARY:
Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) has been the most performed bariatric surgical intervention until a few years ago, due to its good results in terms of weight loss and remission of comorbidities such as hypertension, type 2 diabetes mellitus, dyslipidemia and obstructive sleep apnea syndrome. However, more than 25% of patients do not obtain the expected result.

There is no uniform technique to perform a LRYGB, but traditionally it was constructed using a long alimentary limb (AL) and a short biliopancreatic limb (BPL). There is no current consensus on the ideal length of the LRYGB limbs.

The distal gastric bypass at the expense of a longer biliopancreatic limb (LBPL-GB) could induce more excess of weight loss (EWL%), but with possible protein malnutrition depending on the length of the remaining common limb.

The aim of this study is compare a LBPL-GB (BPL 150cm, AL 70cm) with LAL-GB (BPL 70cm, AL 150cm).

PRIMARY OUTCOME: to evaluate if there are differences in weight loss. SECONDARY OUTCOME: to assess whether there are differences in both groups in remission of the most common comorbidities and in quality of life.

DESIGN: multicenter, prospective, randomized study in blocks (1:1), blinded for the patient and to the surgeon up to the time of intervention, in patients with indication of RYGB for obesity (BMI>35 with associated comorbidity or BMI>40 with or without comorbidity, excluding those of BMI>50). Intervention: LRYGB type 1 (LAL-GB: 150cm ALand 70cm BPL) or type 2 (LBPL-GB: 70cm AL and 150cm BPL).

The expected result is that the patients with LBPL-GB present better EWL%, and higher remission of their comorbidities than the comparison group

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI 35-40 kg/m2 with associated medical problems (Diabetes Mellitus, Hipertension, Dyslipidemia, Obstructive Sleep Apnea Syndrome) or 40-50 kg/m2 with or without associated medical problems, who comply with the regulatory rules for bariatric surgery in Spain (SECO and AEC)

Exclusion Criteria:

* General contraindications to kind of surgery
* BMI > 50 kg/m2
* Known drug or alcohol abuse
* ASA (American Society of Anesthesiology) physical status classification > III
* Inability to follow the procedures of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2024-10-11 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Excess Weight Loss (%EWL) | From baseline to five years after surgery
  The Excess Weight Loss (%EWL) after surgery. (Preoperatory weight in kilograms - current weight in kilograms) / (preoperatory weight in kilograms) x 100

SECONDARY OUTCOMES:
Remission or improvement of Type 2 Diabetes Mellitus | From baseline to five years after surgery
  Remission or improvement of Type 2 Diabetes Mellitus after surgery, according to the Criteria of American Diabetes Association, Spanish Obesity Surgery Society and Spanish Surgeon Association.
  Complete remission: HbA1c < 6% and normalization of fasting blood glucose (100 mg/dl) without medication during one year minimum. Partial remission: HbA1c 6-6.5% and fasting blood glucose between 100 and 125 mg/dl) without medication.
  Prolonged remission: at least 5 years of remission. Improvement HbA1c < 7%, with pharmacological treatment. ADA criteria (American Diabetes Association)
Remission or improvement of Hypertension | From baseline to five years after surgery
  Remission or improvement of Hypertension after surgery, according to the Criteria of the Spanish Obesity Surgery Society and Spanish Surgeon Association.
  Complete remission: blood pressure (BP) <120/80 without medication Partial remission: systolic BP 120-140 mmHg and diastolic BP 80-89 mmHg without medication.
Remission of improvement of Dyslipidemia | From baseline to five years after surgery
  Remission or improvement of Dyslipidemia after surgery, according to the Criteria of the Spanish Obesity Surgery Society and Spanish Surgeon Association.
  Low-density lipoprotein cholesterol (LDLc) < 100 mg/dl, Triglycerides (TG) < 150 mg/dl, total cholesterol < 200 mg/dl, High-density lipoprotein cholesterol (HDLc) > 60 mg/dl.
Remission or improvement of Obstructive Sleep Apnea Syndrome | From baseline to five years after surgery
  Remission or improvement of Obstructive Sleep Apnea Syndrome after surgery, according to the Criteria of the Spanish Obesity Surgery Society and Spanish Surgeon Association.
  Number of apneic-hypopneic episodes/hour, recorded by polysomnography.

OTHER OUTCOMES:
Quality of life after surgery | From baseline to five years after surgery
  Quality of life with the Bariatric Analysis and Reporting Outcome System (B.A.R.O.S) Scale.
  The score range is from 0 to 6 if the patient doesn´t have comorbidities. The result varies depending on the score. Failed=0, regular=0-1.5, good=1.5-3, very good=3-4.5, excellent=4.5-6.
  The score range is from 0 to 9 if the patient has some comorbidities. The result varies depending on the score. Failed=0-1, regular=1-3, good=3-5, very good=5-7, excellent=7-9.
  We will measure it a year and 5 years after surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Juan José Arroyo Martín, Denia, Alicante
  - Esther Mans Muntwyler, Mataró, Barcelona
  - Débora Acín Gándara, Fuenlabrada, Madrid

IPD SHARING:
Plan to Share IPD: No